CLINICAL TRIAL: NCT05042193
Title: A Prospective Cohort Study of Immunoglobulin G (IgG) Dynamics Against SARS-Co
Brief Title: A Prospective Virtual Study to Evaluate the Longevity of IgG Antibodies in Individuals Exposed to COVID-19
Status: Completed | Type: Observational
Sponsor: Everly Health (Industry)
Responsible Party: Sponsor
Other Study IDs: EW-US-4010-0007
Record Dates: First submitted 2021-09-09; First posted 2021-09-13 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unvaccinated SARS-CoV-2 positive: Participants who have tested positive for SARS-CoV-2, both with and without symptoms, who have not been vaccinated
  Interventions: Other: SARS-CoV-2
- Vaccinated: Participants who were vaccinated against SARS-CoV-2
  Interventions: Other: SARS-CoV-2

INTERVENTIONS:
Other: SARS-CoV-2 — Observational

SUMMARY:
The primary objective of this study is to describe the longevity of IgG against SARS-CoV-2 infection or vaccination.

DETAILED DESCRIPTION:
This virtual clinical study will use a prospective design, to evaluate longevity and seroprevalence of IgG against SARS-CoV-2 in approximately 800 patients as measured by Dried Blood Spots via fingerstick using the Everlywell COVID-19 Antibody Test Home Collection Kit. Participants will be followed up to 9 months at 1, 3, 6 and 9 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Willing to provide informed consent prior to participation.
* Cohort 1 (Arm 1) - Positive test results for SARS-CoV-2 virus by an RT-PCR or Antigen test AND not received any COVID-19 vaccine or participated in any COVID-19 vaccine trial
* Cohort 2 (Arm 2) - Received the COVID-19 vaccine

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Individuals with known conditions or treatments associated with immune impairment, such as cancer and chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who have tested positive for SARS-CoV-2 by either RT-PCR or Antigen test for COVID-19 or have received one of the commercially available SARS-CoV-2 vaccines.
Sampling Method: Non-Probability Sample
Enrollment: 1883 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
To describe the longevity and seroprevalence of IgG against SARS-CoV-2 in a cohort of individuals exposed to SARS-CoV-2 | Up to 9 months

SECONDARY OUTCOMES:
To compare the off-kinetics of IgG positivity against SARS-CoV-2, stratified by age, sex, race, ethnicity, infection symptomaticity, initial viral load | Up to 9 months
To compare the off-kinetics of IgG positivity against SARS-CoV-2 by natural infection vs vaccination | Up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bauer, PhD, Principal Investigator — Everly Health
Locations (1):
- Everlywell, Inc, Austin, Texas, United States